CLINICAL TRIAL: NCT04076852
Title: Gilles de la Tourette Syndrome (TS) and Seasonality: a Pilot Study
Brief Title: Gilles de la Tourette Syndrome (TS) and Seasonality
Status: Terminated | Type: Observational
Why Stopped: Satisfactory results, in terms of both clinical and statistical, were achieved.
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Stagionalità TS (PI: M Porta); L3036 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2018-12-29; First posted 2019-09-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2019-08

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Administration of questionnaires — According to clinical practice, the following questionnaires are administered:
  * Y-GTSS
  * Y-BOCS or cY-BOCS

SUMMARY:
This retrospective and prospective observational study intends to evaluate the correlation between seasons and the variation of the syndromic structure of the Tourette.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the Tourette Center since January 2012.
* Males and females.
* Age between 6 and 50 (completed).
* Diagnosis of Tourette syndrome ascertained
* Presence of a value equal to or greater than 15/40 of the Y-BOCS.

Exclusion Criteria:

* Presence of allergic pathology.
* Presence of significant psychiatric symptoms, with the exception of those belonging to the Tourette Syndrome itself (eg ADHD, OCD)

Ages: 6 Years to 50 Years | Sex: All
Age Groups: Child, Adult
Study Population: Being a pilot study it was not possible to develop a sample study, but the sample number is designed based on the tourette center turnout
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Y-GTSS score at 6 months. | 4, 8, 12 months.
  The primary objective is to investigate the correlation between seasons and different phenotypic variation through the administration of a specific questionnaire (Y-GTSS) and questions about the subjective perception of the ticcogenic variation.

SECONDARY OUTCOMES:
Change from baseline Y-BOCS score at 6 months. | 4, 8, 12 months.
  Secondary objective is to investigate the correlation between seasons and variation of severity of obsessive-compulsive disorder (OCD) through the administration of Y-BOCS, a questionnaire indicated to evaluate the severity of obsessive-compulsive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Porta, Principal Investigator — IRCCS Orthopedic Institute Galeazzi
Locations (1):
- IRCCS Galeazzi Hospital, Milan, Lombardy, Italy